CLINICAL TRIAL: NCT03227731
Title: Immediate or Deferred Pre-exposure Prophylaxis for HIV Prevention: Safe Options for Pregnant and Lactating Women An Open-Label Randomised Control Study
Brief Title: Immediate or Deferred Pre-exposure Prophylaxis for HIV Prevention: Safe Options for Pregnant and Lactating Women
Acronym: PrEP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: Centre for the AIDS Programme of Research in South Africa (Network); Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Dhayendre Moodley, PhD, Professor, University of KwaZulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UKwaZulu
Record Dates: First submitted 2017-06-30; First posted 2017-07-24 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: HIV-1-infection
Keywords: Preexposure prophylaxis; safety; HIV prevention; pregnant women; lactating women
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir

STUDY DESIGN:
Intervention Model Description: Pregnant women considered at high risk for HIV infection will be randomized to commencing PrEP in pregnancy with continued use throughout breastfeeding or deferred PrEP until breastfeeding cessation. Women in either group will receive the standard of care for prevention of HIV and other sexually transmitted infections.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Intervention - Truvada) (Active Comparator): Standard HIV Prevention strategy plus a once daily dose of Truvada (FTC 200mg/TDF 300mg tablet) initiated in pregnancy and continuing until cessation of breastfeeding or 18 months postdelivery whichever is earliest and thereafter the option to continue PrEP post breastfeeding cessation.
  Interventions: Drug: Truvada
- Arm B (Control - Standard of Care) (No Intervention): Standard HIV Prevention strategy throughout pregnancy until 18 months postdelivery plus the offer to initiate PrEP post breastfeeding cessation

INTERVENTIONS:
Drug: Truvada — Truvada (Truvada (emtricitabine 200mg/tenofovir disoproxil fumarate 300mg) is in a fixed-dose combination (FDC) tablet formulation and is proven safe for the prevention and treatment of HIV in non-pregnant and non-lactating women.
  Other Names: emtricitabine 200mg/tenofovir disoproxil fumarate 300mg)
  Arms: Arm A (Intervention - Truvada)

SUMMARY:
An Open Label randomized control study. To explore the safety of Truvada when used as PrEP during pregnancy and lactation. Pregnant women considered at risk for HIV infection and willing to participate in this randomized control study will be randomized to commencing PrEP in pregnancy and continued use throughout breastfeeding or deferred PrEP until breastfeeding cessation. All women will receive the standard of care for prevention of HIV and other sexually transmitted infections.

Arm A: (Intervention): Standard HIV Prevention strategy plus a once daily dose of Truvada (FTC 200mg/TDF 300mg tablet) initiated in pregnancy, continuing until cessation of breastfeeding or 18 months postdelivery whichever is earliest and thereafter the option to continue PrEP post breastfeeding cessation.

Arm B: (Control): Standard HIV Prevention strategy throughout pregnancy until cessation of breastfeeding plus the offer to initiate PrEP post breastfeeding cessation.

Standard HIV prevention strategy includes risk reduction counselling, sexually transmitted infection (STI) screening and treatment, condom promotion and inviting the sexual partner to receive HIV counselling and testing (HCT) and referral for antiretroviral therapy (ART) if he tests positive.

Main Outcome Measure: Renal function, pregnancy outcomes, bone health and infant growth.

Other Outcome Measure: Incident HIV infections, adherence to PrEP, drug resistance and mother-to-child transmission of HIV.

DETAILED DESCRIPTION:
Background:

It is becoming increasingly evident that women remain vulnerable to HIV infection during pregnancy and even more so postdelivery. In a meta-analysis, using data from 19 international cohorts, Drake et al concluded that the pooled HIV incidence rate during pregnancy/postpartum was 3.8/100 per woman years (PWY) (95% Confidence Interval (CI) 3.0-4.6): 4.7/100 PWY during pregnancy and 2.9/100 PWY postpartum. In earlier South African studies (2005-2009) investigators reported HIV seroconversion rates ranging from 1.3% to 3.0% in pregnancy [4-6]. Dinh et al in 2010-2012 reaffirmed the high seroconversion rate among pregnant women attending public health facilities in South Africa; 3.3% (95% CI: 2.8%-3.8%) women seroconverted in pregnancy [7]. In an evaluation of PMTCT program indicators in KwaZulu-Natal in 2015 the HIV seroconversion rate among 78 906 pregnant HIV uninfected women was estimated as 1.8% (95%CI 1.0-2.9) in pregnancy and 5% (among 26 455 breastfeeding women) in the postnatal period.

Rationale:

Truvada, an antiretroviral agent containing emtricitabine (200 mg) and tenofovir disoproxil fumarate (300 mg) in a fixed-dose combination (FDC) tablet formulation is widely used in pregnant women as part of a combination treatment regimen and as prophylaxis to prevent mother-to-child transmission of HIV. Truvada is also the drug of choice in PrEP and currently recommended by the World Health Organization (WHO) for people at substantial risk of HIV infection (incidence >3%). Pregnant women were excluded from participating in PrEP trials because of the lack of safety data in pregnancy. Available human and animal data suggest that TRUVADA does not increase the risk of major birth defects overall compared to the background rate and there are limited safety data for TDF/FTC when used in HIV uninfected pregnant women. In the past five years, PrEP trials have explored the use of Tenofovir alone or in combination with Emtricitabine in a once daily regimen, resulting in varying efficacy outcomes that have been largely associated with adherence. Much of the safety data have been generated in studies involving ART in HIV infected pregnant women. The majority of these studies indicate no added adverse effect of TDF on pregnancy outcomes. The few studies of TDF use in HIV uninfected women are treatment studies to prevent mother-to-child transmission of Hepatitis B and only 2 studies of TDF as PrEP use among women who subsequently fell pregnant post enrolment. However, exposure to TDF during pregnancy in these PrEP studies is limited since TDF was halted once pregnancy was diagnosed. Only a handful of studies have demonstrated the excretion of TDF into breastmilk and have concluded that these are relatively low doses of exposure to the infant. When women were given TDF 300mg/FTC 200mg as part of the triple drug regimen in Option B+ program in Malawi the Tenofovir concentrations in breastmilk were very low (breast milk/maternal plasma ratio = 0.08) [59]. Additional studies are needed to explore the effect of long term TDF exposure during breastfeeding on child growth and child health. Considering HIV uninfected women are encouraged to breastfeed for at least a year, studies exploring the long term effect of breastmilk exposure to TDF when used as PrEP in the mother, are needed.

Goal:

To explore the safety of Truvada when used as PrEP in combination with current recommendations for prevention of sexually transmitted infections in young women at substantial risk of HIV acquisition during pregnancy and lactation.

Study Population:

Pregnant women, at their first antenatal visit, HIV uninfected, without evidence of maternal or fetal complications and at risk for HIV infection.

Sample Size:

To compare the frequency and seriousness of adverse events in women receiving tenofovir/emtricitabine in pregnancy as opposed to women not receiving tenofovir/emtricitabine in pregnancy, we have based our sample size on the main clinically relevant pregnancy outcome. Although all pregnancy outcomes will be compared between the intervention (immediate PrEP) and control (deferred PrEP) groups, we based our sample size on the expected preterm delivery proportion among HIV uninfected women (South Africa 18.5%, Botswana 19%). A sample size of 421 in the Immediate PrEP group and 421 in the Deferred PrEP group (i.e. 842 in total) achieves 80% power to detect a non-inferiority margin difference between the group proportions of 0.075 or 7.5%. The reference group proportion (deferred PrEP) of pre-term delivery pregnancy outcome as a main clinically-relevant adverse event is 0.185 or 18.5%.

Study Design: An Open Label randomized control study. Pregnant women considered at high risk for HIV infection will be randomized to commencing PrEP in pregnancy with continued use throughout breastfeeding or deferred PrEP until breastfeeding cessation. Women in either group will receive the standard of care for prevention of HIV and other sexually transmitted infections.

Study Duration:

Mother: From the first antenatal visit in pregnancy until 18 months post-delivery.

Infant: From birth until 18 months of age. Approximately 12 months for planned accrual and 24 months for complete follow-up. The study period is expected to span 3 years.

Study Products:

Truvada (emtricitabine 200mg/tenofovir disoproxil fumarate 300mg) is in a fixed-dose combination (FDC) tablet formulation and is proven safe for the prevention and treatment of HIV in non-pregnant and non-lactating women.

Study Arms:

Arm A: (Intervention) Standard HIV Prevention strategy plus a once daily dose of Truvada (FTC 200mg/TDF 300mg tablet) initiated in pregnancy and continuing until cessation of breastfeeding or 18 months postdelivery whichever is earliest and thereafter the option to continue PrEP post breastfeeding cessation.

Arm B: (Control) Standard HIV Prevention strategy throughout pregnancy until 18 months postdelivery plus the offer to initiate PrEP post breastfeeding cessation.

Primary Objective:

• To compare the frequency and seriousness of specific adverse events related to TDF/FTC in women and their children in Arm A (exposure to TDF/FTC) and Arm B (no exposure to TDF/FTC) during pregnancy until breastfeeding cessation.

Secondary Objectives:

* To estimate HIV incidence in women in Arm A with Arm B at delivery and at 18 months post-delivery.
* To determine the interdependency of adherence to a once daily oral TDF/FTC regimen and standard HIV prevention methods during pregnancy and postdelivery.
* To measure antiretroviral drug (TDF/FTC) level in women and their infants in association with adherence, safety and level of protection (plasma and breastmilk)
* To detect drug resistance among women who acquire HIV infection and correlate the treatment outcomes (after initiating immediate antiretroviral (ARV) treatment) with drug resistance
* To determine mother-to-child transmission of HIV among women who acquire incident infections during pregnancy and breastfeeding and the frequency of drug resistance in their infected babies

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Confirmed HIV-1 uninfected.
* Willing to provide screening informed consent
* Currently pregnant
* Considered high risk for HIV infection

  * Unprotected sex during pregnancy
  * HIV status of current sexual partner is positive or unknown
* Results of Hepatitis B Virus (HBV) screening (HBsAg testing) available from specimen obtained within 30 days prior to entry
* Plans to deliver in the study affiliated hospital
* Has no plans to move residence outside of the catchment area during the 18 months following delivery

Exclusion Criteria:

* HIV infected
* <18 years of age
* The following laboratory values from a specimen obtained within 30 days prior to study entry:

  * Hemoglobin <9.5 g/dL
  * White Blood Cell Count (WBC) < 1500 cells/mm3
  * Absolute Neutrophil Count (ANC) < 750 cells/mm3
  * Platelets < 100,000 cells/mm3
  * Alanine Aminotransferase (ALT) > 2.5 x upper limit of normal (ULN)
  * Estimated creatinine clearance of < 70 ml/min using the cockcroft-gault equation for women: {([140 - age (years)] x [weight (kg)]) ÷ [72 x serum Cr (mg/dL)]} x 0.85
  * Hepatitis B surface antigen (HBsAg) positive
* Participation in any other study
* In labour - at onset or beyond
* Serious illness (including TB) and/or hospitalization
* Receipt of TB treatment within 30 days prior to study entry
* Fetus detected with serious congenital malformation (ultrasound not required to rule out this condition)
* History of documented structural or conduction heart defect
* Social or other circumstances which would hinder long-term follow-up, in the opinion of the site investigator
* Currently incarcerated
* Substance or alcohol abuse (a score of >8 on the WHO Alcohol Use).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 540 (Actual)
Dates: Start 2017-09-28 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy Outcome-Preterm Deliveries | Within 72 hours postdelivery
  Number of preterm deliveries < 37 weeks gestation
Bone Mineral Density in mother and infant | 6 weeks postdelivery, and thereafter 6 monthly until week 74
  Number of participants with decreased bone mineral density of hip and spine
Pregnancy Outcome-Low Birth Weight | Within 72 hours
  Number of Low birth weight babies <2500g

OTHER OUTCOMES:
Incident HIV infection | Monthly during pregnancy and until 74 weeks postdelivery
  Number of Incident HIV infections in women
Adherence to PrEP | Monthly during pregnancy and until 74 weeks postdelivery
  Number of women with >90% adherence to PrEP

CONTACTS AND LOCATIONS:
Overall Officials: Dhayendre Moodley, PhD, Principal Investigator — University of KwaZulu
Locations (1):
- University of KwaZulu-Natal, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khoza N, Desmond AC, Moodley D. Adherence to Oral HIV Pre-exposure Prophylaxis During Pregnancy and the Post-partum Period: Lessons Learned in an Open-Labelled Clinical Trial. AIDS Behav. 2025 Nov 15. doi: 10.1007/s10461-025-04952-z. Online ahead of print. PMID 41240274
- [Derived] Moodley D, Lombard C, Govender V, Naidoo M, Desmond AC, Naidoo K, Mhlongo O, Sebitloane M, Newell ML, Clark R, Rooney JF, Gray G; CAP016 Team. Pregnancy and neonatal safety outcomes of timing of initiation of daily oral tenofovir disoproxil fumarate and emtricitabine pre-exposure prophylaxis for HIV prevention (CAP016): an open-label, randomised, non-inferiority trial. Lancet HIV. 2023 Mar;10(3):e154-e163. doi: 10.1016/S2352-3018(22)00369-1. Epub 2023 Feb 3. PMID 36746169

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/31/NCT03227731/Prot_SAP_ICF_000.pdf